CLINICAL TRIAL: NCT03231670
Title: Analysis of Blood Cells Innate Immune Response in Patients With Lobar Pneumonia
Brief Title: Innate Immune Response of Blood Cells in Patients With Pneumonia
Acronym: ASTRAL
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Institut Pasteur de Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RT-12
Record Dates: First submitted 2017-07-24; First posted 2017-07-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Lobar Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples 5ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lobar pneumonia: Inpatient with lobar pneumonia will undergo a blood sampling during their hospitalization and after resolution of the infection (2 Months)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — 5ml blood will be taken in addition to standard sampling

SUMMARY:
Pulmonary bacterial infections such as exacerbations of chronic bronchitis, nosocomial and community-acquired pneumonia represent a major public health issue. Antibiotics have shown their efficacy by direct antimicrobial activity and their limit particularly in case of multidrug-resistant microorganisms or in treating patients with aggravating pathologies. Innate immunity could be an alternative or complementary therapeutic pathway. Innate immunity receptors bind universal and invariant microbial molecular patterns present in bacteria, virus, fungus or parasite. Toll-like Receptors (TLR) activation by microbial agonist stimulates the innate immunity response which results in the production of chemokines, cytokines, antimicrobial molecules and the recruitment of innate cells.

The " Pulmonary Infection and Innate Immunity " team of the Immunity and Infection Center in Lille (Group of Dr. Sirard and Carnoy) has a long expertise in the study of TLR5 and its agonist, the flagellin, a structural protein of bacterial flagella. TLR5 is expressed on the cell surface of macrophages, monocytes, dendritic and epithelial cells. Several studies in mice have shown the flagellin prophylactic potential during bacterial infections through a TLR5 dependent stimulation of innate immunity. Recently, the group of Dr. Sirard and Carnoy has shown that flagellin can be used in association with antibiotics to treat Streptococcus pneumoniae respiratory infections in mice. The results demonstrate that an agonist of TLR can increase the therapeutic index of an antibiotic and improve the pulmonary anti-infectious reaction. This innovative approach allows us to consider new antibacterial strategies where antibiotics have reached their limit (nosocomial infection, multidrug-resistant bacteria…). TLR agonists can activate multiple human cell type. Indeed, blood cells activation by TLR agonists have been recently characterized in healthy volunteers.

However, there is no available data on the ability of TLR agonists to activate cells from patients with infectious pneumopathies. A study in these patients is inevitable if one is to consider the therapeutic use of agonists in respiratory pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized in the department of pneumology for whom clinical, radiological and biological criteria confirm the diagnosis of lobar pneumonia
* Beneficiary of the French National Health Insurance Fund
* Signed informed consent form

Exclusion Criteria:

* Patient under guardianship
* Patient with acute respiratory distress syndrome or septic shock
* Pregnant women
* Patient with HIV, HCV or Mycobacterium tuberculosis
* Transplanted patient receiving immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient hospitalized in the department of pneumology for whom clinical, radiological and biological criteria confirm the diagnosis of lobar pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Change in IL-6 specific transcripts | Baseline and 2 months
  IL-6 specific transcripts will be measured in blood mononuclear cells after stimulation with a TLR5 agonist.

SECONDARY OUTCOMES:
Change in expression of innate immunity genes after stimulation by TLR2 agonist | Baseline and 2 months
Change in expression of innate immunity genes after stimulation by TLR4 agonist | Baseline and 2 months
Change in expression of innate immunity genes after stimulation by TLR5 agonist | Baseline and 2 months
Change in expression of innate immunity genes after stimulation by TLR9 agonist | Baseline and 2 months
Change in ELISA assay on mediators of inflammation with stimulation by TRL2 agonist | Baseline and 2 months
  ELISA assay on mediators of inflammation in the supernatant of blood mononuclear cells stimulated by TRL2 agonist
Change in ELISA assay on mediators of inflammation with stimulation by TRL4 agonist | Baseline and 2 months
  ELISA assay on mediators of inflammation in the supernatant of blood mononuclear cells stimulated by TRL4 agonist
Change in ELISA assay on mediators of inflammation with stimulation by TRL5 agonist | Baseline and 2 months
  ELISA assay on mediators of inflammation in the supernatant of blood mononuclear cells stimulated by TRL5 agonist
Change in ELISA assay on mediators of inflammation with stimulation by TRL9 agonist | Baseline and 2 months
  ELISA assay on mediators of inflammation in the supernatant of blood mononuclear cells stimulated by TRL9 agonist
Genotyping of TLR 2 gene | Baseline
Genotyping of TLR 4 gene | Baseline
Genotyping of TLR 5 gene | Baseline
Genotyping of TLR 9 gene | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Carnoy, PhD, Study Director — Institut Pasteur de Lille; Jean-Claude Sirard, PhD, Study Director — Institut Pasteur de Lille
Locations (1):
- Hôpital Saint-Philibert, Lomme, Hauts-de-France, France